CLINICAL TRIAL: NCT02036268
Title: A Prospective, Single-Center Study to Assess the Impact of Pre- and Post-Surgical Ostomy Care Education on Patient Outcomes and Quality of Life
Brief Title: Different Levels of Patient Education for Care of Ostomy Site
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of study coordinator and time.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Bruce W. Robb, Clinical Associate Professor of Surgery, Indiana University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1202007926
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Ostomy
Keywords: Ostomy education; Education; care of ostomy site

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard (Active Comparator): Subjects will receive standard ostomy education.
  Interventions: Behavioral: Standard
- Pre-Operative Education (Experimental): In addition to standard ostomy education, subjects will receive additional education pre-operatively.
  Interventions: Behavioral: Standard; Behavioral: Pre-operative Education
- Two-week Post Operative Education (Experimental): In addition to standard ostomy education, subjects will receive additional education two weeks following surgery.
  Interventions: Behavioral: Standard; Behavioral: Pre-operative Education; Behavioral: Two-week Post Operative Education

INTERVENTIONS:
Behavioral: Standard — Standard ostomy education
Behavioral: Pre-operative Education — In addition to standard ostomy education, an additional pre-operative ostomy education session will be conducted with the subject.
  Arms: Pre-Operative Education; Two-week Post Operative Education
Behavioral: Two-week Post Operative Education — In addition to standard ostomy education and an additional pre-operative ostomy education session, another ostomy education session will be conducted with the subject two weeks post-op.
  Arms: Two-week Post Operative Education

SUMMARY:
This is a randomized study of standard versus extra ostomy education.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of pre-operative and post-operative ostomy education compared to standard of care ostomy education.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years of age at the time of consent.
* Scheduled to undergo surgery at IU Health North Hospital that will results in a temporary or permanent colostomy or ileostomy for a benign or malignant disease process.
* Are willing and able to provide written informed consent for participation in the study and authorization for release of health information.
* Are willing and able to attend up to two additional clinic visits at IU Health North Hospital for the purpose of ostomy teaching and care.
* Subjects who currently do NOT have a urostomy or any other type of urinary diversion and/or are NOT planning to have a urostomy or any other type of urinary diversion as part of the surgery procedures at the time of their surgery for placement of colostomy or ileostomy.
* Subjects who do NOT have any history of prior colostomy or ileostomy.

Exclusion Criteria:

* Subjects not meeting any of the above eligibility criteria.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-05; Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Stoma Quality of Life Scale (SQOLS) | Six weeks
  The SQOLS assesses patient quality of life on a 5-point Likert type scale, where 1 = Never and 5 = Always. Higher scores indicate a greater self-reported quality of life.

SECONDARY OUTCOMES:
Skin integrity at the ostomy site by lesion type | Six weeks
  Skin integrity will be assessed by the SACS Instrument (Studio Alterazioni Cutanee Stomali). The SACS classifies lesion type.
Skin integrity at the ostomy site by location | Six weeks
  Skin integrity will be assessed by the SACS Instrument (Studio Alterazioni Cutanee Stomali). The SACS classifies lesion location.
Number of appliance changes | Six weeks
  Subjects will be asked to record the number of wafer and/or bag changes completed during study participation in a patient diary.
Stoma Care Self-Efficacy Scale (SCSES) | Six weeks
  The SCSES assesses patient quality of life on a 4-point Likert type scale, where 1 = Not At All and 5 = Almost Always. Higher scores indicate a greater self-reported quality of life related to self-confidence in stoma care.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce W Robb, MD, Principal Investigator — Indiana University, Department of Surgery
Locations (1):
- Indiana University Health North Hospital, Carmel, Indiana, United States

IPD SHARING:
Plan to Share IPD: No